CLINICAL TRIAL: NCT01919866
Title: Haploidentical Stem Cell Transplantation With CD3/CD19 Depleted Stem Cells in Pediatric Patients With Refractory Hematological and Oncological Diseases
Brief Title: Safety Study of CD3/CD19 Depleted Haploidentical Stem Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Children's Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Peter Lang, Prof. Dr. med., University Children's Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1075/01 PEI
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Acute Leukemias; Aplastic Anemia; Childhood Solid Tumor
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplantation of CD3/CD19 depleted stem cells (Experimental): Patients receive a minimum dosage of 10x10E6/kg bodyweight CD3/CD19 depleted CD34+ stem cells. Maximum dosage of residual T cells will be 1x10E5/kg BW
  Interventions: Other: Transplantation of CD3/CD19 depleted stem cells

INTERVENTIONS:
Other: Transplantation of CD3/CD19 depleted stem cells

SUMMARY:
Feasibility and toxicity of haploidentical transplantation of CD3/CD19 depleted stem cells in combination with a toxicity reduced conditioning regimen or with standard conditioning regimens according to underlying disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with primary refractory or relapsed disease (including relapse after previous SCT and active disease)
* AML in complete remission of refractory
* MDS RAEB-t/secondary AML
* ALL
* CML
* Non-Hodgkin Lymphoma / Hodgkin Lymphoma
* non malignant diseases (aplastic anemia, thalassemia, SCID)
* relapsed Neuroblastoma
* relapsed soft tissue sarcoma (Rhabdomyosarcoma, Ewing sarcoma, PNET
* soft tissue sarcoma with primary bone metastases or bone marrow
* in whom no matched donor was available,

Exclusion Criteria:

* < 6 months after previous HSCT
* active cerebral seizure conditions
* massive progression of leukemias or solid tumours before planned trp.
* left ventricular ejection fraction <25%
* creatinine clearance <40ml/min before conditioning
* respiratory insufficiency with oxygen demand or DLCO <30%
* Bilirubin >4mg/dl, GOT/GPT >400
* severe infection (HIV, Aspergillosis)
* pregnancy

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Engraftment rate and transplant related mortality | 365 days
  engraftment rate will be evaluated by leukocyte counts in peripheral blood . Definition of engraftment: >500 neutrophiles/µl blood. Transplant related mortality will be evaluated at day 100 and day 365 post transplant

SECONDARY OUTCOMES:
Graft versus Host disease and speed of immune reconstitution | 365 days
  Incidence of acute and chronic GvHD will be evaluated according to Glucksberg criteria. Immune recovery will be evaluated by flow cytometry. Percentages and numbers of T, B and NK cells will be measured weekly until day 100, afterwards on day 180 and 365.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lang, MD, Principal Investigator — University Children's Hospital Tuebingen
Locations (5):
- University Children's Hospital, Graz, Austria
- Germany (4):
  - University Children's Hospital, Halle
  - Medizinische Hochschule Zentrum für Kinderheilkunde, Hanover
  - University Children's Hospital, Jena
  - University Children's Hospital, Tübingen